CLINICAL TRIAL: NCT07192055
Title: Self-sampling to Optimize Anal Lesion Outcomes (SOLO)
Brief Title: Self-sampling to Optimize Anal Lesion Outcomes
Acronym: SOLO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: National Cancer Institute (NCI) (NIH); University of Chicago (Other); Froedtert Hospital (Other); M.D. Anderson Cancer Center (Other)
Responsible Party: Principal Investigator, Alan Nyitray, PhD, Associate Professor, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: PRO00054186; R01CA298844 (NIH)
Record Dates: First submitted 2025-09-10; First posted 2025-09-25 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Anal Cancer
Keywords: anal cancer; human papillomavirus
MeSH Terms: conditions — Anus Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: When care providers are scheduling cytology appointments, they will not know the participant arm assignment. When specimens are sent to laboratories, the lab will not know the participant arm assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Self-sampling (Experimental): Participants will self-sample the anal canal with a swab. They will do this at home and at a clinic.
  Interventions: Other: Nylon-flocked Swab
- Clinician sampling (Active Comparator): A clinician will collect a sample from the anal canal of the participant with a swab. They will do this at the clinic.
  Interventions: Behavioral: Self-sampling; Other: Nylon-flocked Swab
- Nylon-flocked swab (Experimental): This is a swab with nylon-flocked material at the tip.
  Interventions: Behavioral: Self-sampling
- Dacron swab (Active Comparator): This is a swab with a Dacron tip.
  Interventions: Behavioral: Self-sampling; Other: Nylon-flocked Swab

INTERVENTIONS:
Behavioral: Self-sampling — Self-sampling instructions will be provided to participants who will insert the swab into the anus to collect cells. Then the participant will put the swab in a vial of transport fluid for assessment at a laboratory.
  Other Names: self-collection
  Arms: Clinician sampling; Dacron swab; Nylon-flocked swab
Other: Nylon-flocked Swab — At the cytology appointment, participants may receive self-sampling or clinician sampling with 1 of 2 kinds of swabs. The nylon-flocked swab is the intervention and will be assessed on patient acceptability and patient and clinician ability to collect an adequate sample.
  Arms: Clinician sampling; Dacron swab; Self-sampling

SUMMARY:
The purpose of this research study is to find ways to increase anal cancer screening among people at increased risk for anal cancer. This study will try to find out if persons will do an intervention (self-sampling of the anal canal) and if it affects cytology and high-resolution anoscopy (HRA) appointment attendance. Secondarily, the study will assess if a person who gets their choice of either self-sampling or healthcare provider sampling affects clinic attendance.

ELIGIBILITY:
A potential study subject who meets all of the following inclusion criteria is eligible to participate in the study. Note that these criteria apply regardless of HPV vaccination status or disability status.

Inclusion Criteria:

1. Age ≥ 35 years for those who are HIV-positive or ≥ 45 years for those who are HIV-negative.
2. Must be either:

   1. A cisgender or transgender sexual minority man, or
   2. A transgender woman who has sex with men.
3. Resides in Chicago, Houston, or Milwaukee metropolitan area.
4. Is willing to attend a study clinic.
5. Speak and understand either English or Spanish
6. Ability to understand a written informed consent document, and the willingness to sign it.

Exclusion Criteria:

A potential study subject who meets any of the following exclusion criteria is ineligible to participate in the study.

1. Was a participant in the PAC Self-Swab Study in Milwaukee.
2. Currently on anticoagulants, with the exception of aspirin or non-steroidal anti-inflammatory drugs (NSAIDs), e.g., ibuprofen, naproxen.
3. Diagnosed with hemophilia, cirrhosis with bleeding varices, or thrombocytopenia.
4. Presence of any contraindicating severe disease or condition, e.g., anal stenosis.
5. Plans to move within 12 months after enrollment.

Min Age: 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — cisgender males and transgender persons who have sex with men
Enrollment: 572 (Estimated)
Dates: Start 2025-11-18 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
Effect of the self-sampling intervention at cytology | 1 month
  Determine the number of individuals who attend the cytology appointment after exposure to the self-sampling intervention.
Effect of self-sampling intervention at high-resolution anoscopy | 2 months
  Determine the number of individuals who attend the high-resolution anoscopy appointment after exposure to the self-sampling intervention.

SECONDARY OUTCOMES:
Effect of the self-sampling intervention at cytology on people with human immunodeficiency virus (HIV) | 1 month
  Determine the number of individuals with HIV who attend the cytology appointment after exposure to the self-sampling intervention.
Effect of the self-sampling intervention at high-resolution anoscopy on people with HIV | 2 months
  Determine the number of individuals with HIV who attend the high-resolution anoscopy appointment after exposure to the self-sampling intervention.
Effect of the self-sampling intervention at cytology on people randomized to their preferred sampling method | 1 month
  Assess the number of participants who attend their cytology appointment in the group randomized to their preferred sampling method.
Effect of the self-sampling intervention at high-resolution anoscopy on people randomized to their preferred sampling method | 2 months
  Assess the number of participants who attend their high-resolution anoscopy appointment in the group randomized to their preferred sampling method.

OTHER OUTCOMES:
Effect of the self-sampling intervention among Black individuals at cytology | 1 month
  Determine the number of Black individuals who attend the cytology appointment after exposure to the self-sampling intervention.
Effect of the self-sampling intervention among Black individuals at high-resolution anoscopy | 2 months
  Determine the number of Black individuals who attend high-resolution anoscopy appointments after exposure to the self-sampling intervention.
Assess the adequacy of nylon-flocked swabs | 1 month
  Determine the number of nylon-flocked swabs that are cytologically adequate (defined as 2000-3000 nucleated squamous cells/mm3).
Assess the adequacy of Dacron swabs | 1 month
  Determine the number of Dacron swabs that are cytologically adequate (defined as 2000-3000 nucleated squamous cells/mm3).
Assess participant pain after using the nylon-flocked swab | 1 month
  The Wong-Baker FACES® Pain Rating Scale measures the severity of pain, if any. Possible scores range from 0 to 10 with higher scores indicating increased severity of pain.
Assess participant pain after using the Dacron swab | 1 month
  The Wong-Baker FACES® Pain Rating Scale measures the severity of pain, if any. Possible scores range from 0 to 10 with higher scores indicating increased severity of pain.
Assess participant comfort after using the nylon-flocked swab | 1 month
  The variable comfort measures the individual's reported comfort on a 4-point Likert scale from Strongly Agree to Strongly Disagree. Possible scores range from 1 to 4 with higher scores indicating decreased comfort after using the nylon-flocked swab.
Assess participant comfort after using the Dacron swab | 1 month
  The variable comfort measures the individual's reported comfort on a 4-point Likert scale from Strongly Agree to Strongly Disagree. Possible scores range from 1 to 4 with higher scores indicating decreased comfort after using the Dacron swab

CONTACTS AND LOCATIONS:
Overall Officials: Alan Nyitray, PhD, Principal Investigator — Medical College of Wisconsin
Locations (3):
- United States (3):
  - University of Chicago, Chicago, Illinois
  - The University of Texas M.D. Anderson Cancer Center, Houston, Texas
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Fully de-identified datasets will be shared with properly trained investigators after assessment of institutional policies, Medical College of Wisconsin Human Protections Committee rules, as well as local, state, and Federal laws and regulations.
Time Frame: Data will become available one year after study completion.
Access Criteria: Fully de-identified datasets will be shared with properly trained investigators after assessment of institutional policies, Medical College of Wisconsin Human Protections Committee rules, as well as local, state, and Federal laws and regulations.